CLINICAL TRIAL: NCT00170586
Title: Novel Protective Underglove
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 03-241; PHS 2002-2
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2007-03

CONDITIONS: Bacterial Diseases
Keywords: Underglove, polyvinylidene fluoride, acrylic polymer
MeSH Terms: conditions — Bacterial Infections

INTERVENTIONS:
Device: Underglove coating (skin barrier)

SUMMARY:
Bloodborne pathogens are infectious bacteria, viruses, or other disease-causing germs carried in blood or other body fluids. These germs include hepatitis B and C viruses and HIV. Surgical and examination gloves are worn by health care workers to reduce the risk of workers catching germs from patients or patients catching germs from workers. The purpose of this study is to further develop polyvinylidene fluoride coatings for use as a protective coating worn underneath the gloves. Some health care workers may have tiny cuts on their hands that need to be protected, and gloves can have defects such as tiny holes that can allow germs to travel through them. The undercoating can add an additional layer of protection under gloves. The coating is applied in liquid form to hands and dries as a film without wrinkling, tearing, lifting, or bubbling. The liquid contains chemicals that fight germs. The coating also provides protection from skin irritation caused by the latex in some gloves.

DETAILED DESCRIPTION:
The goal of this project is to complete development of a unique thin film technology to be used as a skin barrier underneath surgical and examination gloves. The technology, which is antimicrobial upon application to skin, has been developed to reduce transmission of bacteria and bloodborne pathogens, and is expected to protect skin from the detrimental effects of chronic glove occlusion and hand washing. Due to the increased prevalence of human immunodeficiency virus (HIV) and hepatitis, the efficacy of surgical and examination gloves has become an important safety issue, especially for health care workers where occupational exposure to pathogens in blood or other body fluids is common. Transmission can occur from both caregiver to patient, and from patient to caregiver. However, glove leaks are frequent and the potential for pathogen transmission is of great concern. In addition, as awareness of the hazards from bloodborne pathogen transmission increased along with AIDS awareness in the 1990s, the concomitant increased use of disposable gloves has adversely affected skin condition, causing increased cumulative irritation contact dermatitis and heightened dermal sensitization to natural rubber latex. This unique thin film technology is a blend of polyvinylidene fluoride (PVDF) and acrylic polymers that forms thin membrane coatings that provide a tough, flexible barrier to liquids, yet have a "breathable" microporous structure. PVDF-based coatings are applied as a fast drying liquid solution that casts an adherent contiguous film directly on the skin upon drying. The liquid solution is antimicrobial on contact, and after drying, the coatings are durable, resistant to penetration by pathogens, and stay intact for 8 hours or longer. Phase I studies established the feasibility of using the PVDF technology as a protective barrier to be worn underneath gloves. The Phase I studies focused on exploiting the coating's inherent hydrophobicity to create a barrier to bacterial and viral penetration while maintaining breathability and comfort. The coatings demonstrated barrier function to viral and bacterial pathogens in vitro, proved to be safe in animal safety studies, and were shown to be a barrier to liquid in human trials. Phase II studies will complete the development of the PVDF technology for use as a novel protective underglove. The following aims have been designed to demonstrate safety and efficacy of the product and to satisfy Food and Drug Administration (FDA) requirements: implement Good Manufacturing Practices (GMP) and establish packaging; evaluate coating formulations in human subjects for effects on skin physiology; and demonstrate safety of coatings in human studies. A skin coating to be worn under gloves that is antimicrobial on contact, provides a barrier to bloodborne and bacterial pathogens, is a barrier to latex proteins, and could improve skin conditions on hands, would be beneficial to healthcare in the workplace and likewise have significant commercial potential.

ELIGIBILITY:
Inclusion Criteria:

Aim 2a. and Aim 2b1. and Aim 2b2.

1. greater than 18 years of age;
2. healthy subjects as determined by brief medical history;
3. skin in the test area must be devoid of tattoos, scars, moles, vitiligo, keloids, or breaks in the skin;
4. capable of reading, understanding and signing the consent form.

Aim 3.

1. Males/females, 18-70 years of age;
2. healthy subjects as determined by medical history;
3. capable of reading, understanding and signing the consent form.

Aim 2.

1. 18-72 years of age;
2. healthy subjects as determined by a brief medical history;
3. capable of reading, understanding and signing the consent form;
4. skin in the test area must be devoid of tattoos, scars, moles, vitiligo, keloids, or breaks in the skin.

Exclusion Criteria:

Aim 2a. and Aim 2b1. and Aim 2b2. and Aim 2.

1. history or current evidence of a chronic or infectious skin disease
2. pregnant or lactating females. Participating female subjects must agree to use adequate contraceptive measures during the trial. Before entering the study, women of childbearing age will be tested for pregnancy.

Aim 3.

1) active, clinically significant skin diseases such as eczema, atopic dermatitis, psoriasis and skin cancer; 2) severe, chronic asthma; 3) insulin dependent diabetes mellitus or hyperthyroidism (metabolic diseases); 4) routine use of anti-inflammatory medications (i.e., aspirin, ibuprofen, corticosteroids, immunosuppressive drugs or anti-histamines; 5) use of topical drugs at test sites; 6) immunological disorders such as HIV positive, AIDS or systemic lupus erythematosus; 7) participation in any patch test for cumulative irritation or sensitization within the last four weeks; 8) women who are pregnant, lactating, or planning to become pregnant within the next six weeks; 9) mastectomy for cancer involving removal of the lymph nodes; 10) allergy to tapes; 11) subject who has damaged skin in or around test sites which include sunburn, uneven skin tones, tattoos, scars or other disfiguration of the test site; 12) subject who has a condition or is taking or had taken a medication which, in the Investigator's judgement, makes the subject ineligible or places the subject at undue risk; 13) subject who has sensitivity to any of the ingredients in the test articles.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 325
Dates: Start 2003-09; Study Completion 2005-08

CONTACTS AND LOCATIONS:
Locations (1):
- Biomedical Development Corporation, San Antonio, Texas, United States